CLINICAL TRIAL: NCT04922515
Title: Pancreatic Ductal Adenocarcinoma - Microbiome as Predictor of Subtypes
Acronym: PDA-MAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Albrecht Neesse, https://gastroenterologie.umg.eu/ueber-uns/team/neesse/, University Medical Center Goettingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PDA-MAPS
Record Dates: First submitted 2021-05-31; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Oral and rectal swabs for microbiome sequencing — Oral swabs and rectal swabs are collected non-invasively.

SUMMARY:
The prospective clinical trial "PDA-MAPS - Pancreatic ductal adenocarcinoma - Microbiome as Predictor of Subtypes" aims to investigate the prognostic and predictive power of the orointestinal and tumoral microbiome in PDAC patients and associate findings with genetic, transcriptional and clinical data, in particular with treatment response.

DETAILED DESCRIPTION:
The prospective clinical trial "PDA-MAPS - Pancreatic ductal adenocarcinoma - Microbiome as Predictor of Subtypes" aims to investigate the prognostic and predictive power of the orointestinal and tumoral microbiome in PDAC patients and associate findings with genetic, transcriptional and clinical data, in particular with treatment response. Patients with histologically confirmed PDA are enrolled at primary diagnosis and prior to oncological or surgical treatment. Rectal and buccal microbiome swabs as well as detailed clinical records are obtained from all patients. Following DNA extraction, both 16S rRNA and metagenomic sequencing will be performed using ONT sequencing platform. All data and clinical records are centrally stored, visualized and integrated via tranSMART and SEEK platforms.

ELIGIBILITY:
Inclusion Criteria:

- Patients with pancreatic mass suspicious of pancreatic ductal adenocarcinoma

Exclusion Criteria:

* < 18 years
* patients that cannot give informed consent
* pregnant and breastfeeding women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-04-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12 months upon study enrollment
  Progression free survival of patients measured in months

SECONDARY OUTCOMES:
Molecular subtypes of pancreatic cancer | within 3 months of histological diagnosis
  Basal and classical subtype via RNAseq from tissue samples
Response to chemotherapy | up to 6 months after start of therapy
  reponse, partial response and progress according to RECIST within 6 months of therapy initiation

CONTACTS AND LOCATIONS:
Overall Officials: Albrecht Neesse, MD, PhD, Principal Investigator — University Medicine Goettingen
Locations (2):
- Germany (2):
  - University Medical Centre Goettingen, Göttingen
  - University Medical Centre Göttingen, Göttingen

IPD SHARING:
Plan to Share IPD: Undecided